CLINICAL TRIAL: NCT04313309
Title: Evaluating Outcomes of a Integrative Yoga Therapy for People With Chronic Pain
Brief Title: Evaluating Chronic Pain Management Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU021
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Support Group (Experimental): This is the only group in the study consisting of patients with chronic musculoskeletal pain who are receiving the Integrative Yoga Therapy Program
  Interventions: Other: Integrative Yoga Therapy

INTERVENTIONS:
Other: Integrative Yoga Therapy — Individualised intervention developed, consists of a six one to one sessions with patients, followed by home self practiced sessions. The intervention includes yoga movements, yoga breathing, relaxation techniques, reasoning, and other techniques designed to enhance awareness and acceptance of the psychological factors underlying the chronic pain problem.

SUMMARY:
This interventional study seeks to evaluate the overall outcomes of a novel, integrated yoga based intervention for people with chronic musculoskeletal pain and assess the experience of patient to the self care using yoga practices.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic musculoskeletal pain, not accounted for by disease or underlying pathology
* Self referred or referred willing to give informed consent

Exclusion Criteria:

* Autoimmune disorder
* Malignancies
* Cognitively impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Severity of pain and its impact on functioning: Brief Pain Inventory | From baseline to 6-week post intervention
  Brief Pain Inventory

SECONDARY OUTCOMES:
General Quality of Life: Nottingham Health Profile | From baseline to 6-week post intervention
  Nottingham Health Profile
Pain Service Satisfaction: The Pain Service Satisfaction Test (PSST) | From baseline to 6-week post intervention
  The Pain Service Satisfaction Test (PSST)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Chair — Aarogyam UK

IPD SHARING:
Plan to Share IPD: Undecided